CLINICAL TRIAL: NCT02669095
Title: Clinical Evaluation of Approved and Investigational Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-5796
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Visual Disorder
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Test Lens) (Experimental): Subjects will be dispensed the Investigational Contact Lenses (Test) to be worn as daily wear.
  Interventions: Device: Investigational Contact Lenses (Test)
- Arm 2 (Control Lens) (Active Comparator): Subjects will be dispensed the Marketed Contact Lenses (Control) to be worn as daily wear.
  Interventions: Device: Marketed Contact Lenses (Control)

INTERVENTIONS:
Device: Investigational Contact Lenses (Test)
  Other Names: senofilcon C
  Arms: Arm 1 (Test Lens)
Device: Marketed Contact Lenses (Control)
  Other Names: comfilcon A
  Arms: Arm 2 (Control Lens)

SUMMARY:
This study is a multi-site, 5-visit dispensing, bilateral double-arm parallel group design, double-masked clinical trial using an investigational contact lens and a marketed contact lens. The objective is to evaluate comfort of the contact lenses when worn on a daily wear modality.

ELIGIBILITY:
Inclusion Criteria:

* The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must be between 18 to 40 years of age at the time of consent.
* The subject's vertexed spherical equivalent distance refraction must be in the range of +8.00 to -12.00 in each eye.
* Subject wears habitual contact lenses a minimum of 4 days per week, eight hours per day.
* The subject must have best corrected visual acuity of 20/30 or better in each eye.
* The subject must be a habitual frequent replacement daily wear spherical silicone hydrogel soft contact lens wearer in both eyes.
* The subject must be able to wear contact lenses for a minimum of 8 hours each day during the study.
* The subject must have normal eyes (i.e., no ocular medications or infections of any type).

Exclusion Criteria:

* Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
* Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
* Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear.
* Any known sensitive/allergic to Ingredients of OPTI-FREE® PureMoist® solution.
* Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion.
* Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), etc.).
* Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Golden Family Eyecare, Sarasota, Florida
  - Eye Associates of Winter Park, Winter Park, Florida
  - Pickens Family Eye Care, Pickens, South Carolina
  - Total Eye Care PA, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 150 subjects were enrolled in this study. All subjects enrolled into the study were dispensed a study lens. Of the dispensed subjects 146 completed the study and 4 subjects were discontinued.
Groups:
- Senofilcon C: Subjects that were randomized to receive the senofilcon C lens throughout the entire duration of the study.
- Comfilcon A: Subjects that were randomized to receive the comfilcon A lens throughout the entire duration of the study.
Period: Overall Study
Arm/Group | Senofilcon C | Comfilcon A
Started | 75 | 75
Completed | 74 | 72
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Unsatisfactory Lens Fitting | 0 | 1
Not completed — Torn Lens | 0 | 1
Not completed — Visit 5 assessments not completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed a study lens.
Groups:
- Total: Total of all reporting groups
Arm/Group | Senofilcon C | Comfilcon A | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.2 (6.05) | 30.2 (5.62) | 29.2 (5.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 61 | 116
  Male | 20 | 14 | 34
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 2 | 2 | 4
  Black or African American | 12 | 7 | 19
  White | 61 | 65 | 126
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: Participants]
  North America | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Acceptable Lens Fitting
Description: Lens fit was assessed and recorded for each subject and eye at post lens fitting, 1-, 2-, 3- and 4- week follow-up evaluations. Lens fit was a binary response acceptable and unacceptable lens fit. The proportion of eyes with acceptable lens fitting at post lens fit and across all four follow-ups was combined and reported.
Time Frame: Up to 4 Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Proportion of eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Senofilcon C | Comfilcon A
Number analyzed (Participants) | 74 | 72
Number analyzed (Subject Eyes) | 740 | 720
Proportion of eyes | 1 | 0.99

2. Primary Outcome: Overall Comfort
Description: Clue comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. CLUE Comfort was assessed at 1-, 2-, 3 and 4- week Follow-up evaluations. The average CLUE comfort score for each lens was reported for each visit.
Time Frame: Up to 4 Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Senofilcon C | Comfilcon A
Number analyzed (Participants) | 74 | 72
Units on a scale
  1-Week Follow-up | 71.75 (22.193) | 56.68 (27.747)
  2-Week Follow-up | 70.58 (22.500) | 54.69 (30.268)
  3-Week Follow-up | 68.75 (26.108) | 53.43 (29.912)
  4-Week Follow-up | 68.25 (27.137) | 54.57 (30.522)

ADVERSE EVENTS:
Arm/Group | Senofilcon C | Comfilcon A
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days